CLINICAL TRIAL: NCT05025358
Title: A Phase I Study on Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of LP-118 in Patients With Advanced Malignancies
Brief Title: A Study of LP-118 in Patients With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Lupeng Pharmaceutical Company LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-118-CN101
Record Dates: First submitted 2021-07-30; First posted 2021-08-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LP-118 (Experimental): The classic "3+3" design at dose levels of 50mg, 100mg, 200mg, 300mg, 400mg and 500mg will be implemented in this study.
  Interventions: Drug: LP-118 tablet

INTERVENTIONS:
Drug: LP-118 tablet — Subjects will administered orally with LP-118 tablet at the designated dose once daily, using approximately 240 mL of water during a meal or within 30 minutes after a meal, 28 days per cycle. The treatment will continue until progressive disease, unacceptable toxicity, etc.
  Other Names: NWP-4-76

SUMMARY:
This is a phase I, multi-center, open-label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics and clinical activity of LP-118 in patients with advanced malignancies, including solid tumors and lymphomas. LP-118 is a BCL-2/BCL-XL small molecule inhibitor.

DETAILED DESCRIPTION:
LP-118 is an oral selective BCL-2 inhibitor with tuned BCL-XL activity, aiming to improve antitumor efficacy and reduce the risk of thrombocytopenia. Clinical development of LP-118 includes targeting of relapsed or refractory hematological malignancies and solid tumors. This is a multi-center, open-label, Phase 1 dose escalation study of LP-118 in patients with advanced malignancies, including advanced/metastatic solid tumors and relapsed/refractory B cell, T/NK cell lymphomas, to determine the safety, tolerability, pharmacokinetics profile and preliminary anti-tumor efficacy. Upon completion of the Phase 1 dose escalation study and establishment of maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D), the dose expansion study will be implemented in patients with protocol designated type of disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed malignancy, including either of the following disease: relapsed or refractory lymphomas with at least one measurable disease based on Lugano 2014 criteria; or advanced or metastatic solid tumors based on RECIST V1.1 criteria.
* Subjects have a life expectancy of ≥12 weeks, and Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 1.
* Subjects must have adequate bone marrow function independent of blood transfusion or growth factor support per local laboratory reference range at Screening.
* Subjects must have adequate coagulation, renal, and hepatic function, per local laboratory reference range at Screening.
* All acute toxicity from previous anti-tumor treatment or surgery has been alleviated to NCI CTCAE 5.0 ≤ Grade 1.
* All enrolled subjects should take medically approved contraceptives during the entire treatment period and within 90 days after the end of treatment.
* Volunteer and sign informed consent, willing to follow trial protocol.

Exclusion Criteria:

* Subjects who have undergone allogeneic or autologous hematopoietic stem cell transplantation or CAR-T cell therapy (except for lymphoma patients who had received autologous stem cell transplantation or CAR-T cell therapy before 90 days of the first dose of LP-118).
* Subjects who have received the following treatments within 4 weeks or 5 half-lives before the first dose of study drug:

  * Antitumor therapies including myelosuppressive chemotherapy, targeted therapy, biological therapy and/or immunotherapy;
  * Any investigational treatment;
  * Patients who have undergone major surgery, severe trauma or radiotherapy.
* Subjects who have received the following treatments within 1 week before the first dose of study drug:

  * Steroids or traditional herbal medicine for antitumor purposes;
  * Strong and moderate CYP3A inhibitors and inducers, grapefruit and grapefruit juice;
  * Any medications that can cause QTc interval prolongation or torsional tachycardia.
* Solid tumor patients with ITP or AIHA.
* Subjects with known bleeding disease or with a history of non-chemotherapy induced thrombocytopenic bleeding or ineffective platelet transfusion within 1 year before the first dose of study drug.
* Subjects with uncontrollable or CTCAE ≥ grade 2 gastrointestinal bleeding occurred within 90 days before the first dose of study drug.
* Subjects have received the therapeutic dose of anticoagulant or antiplatelet drugs within 1 week before the first dose of study drug.
* Subjects have any serious and/or uncontrolled systemic disease.
* Subjects have poor cardiovascular function, in line with New York Heart Association (NYHA) cardiac function classification ≥ 2 or QTcF greater than 450ms (male) or 470ms (female) on ≥ 3 independent ECG.
* Subjects have disease states where clinical manifestations may be difficult to control, including but not limited to HIV, HBV, HCV, syphilis positive or active bacterial and fungal infections.
* Lymphoma with primary central nervous system (CNS) malignancy or any disease affects the CNS.
* Any gastrointestinal conditions that may severely affect the study drug absorption or pharmacokinetic parameters.
* Subjects who have known severe allergies to study drugs or any excipients.
* Subjects who have evidence of a second primary tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 24 months
  The highest dose that does not cause unacceptable side effects or overt toxicities which will be assessed by NCI CTCAE v5.0.
Adverse events | Up to 24 months
  The incidence and severity of adverse events as assessed by NCI CTCAE v5.0.
Recommended phase II dose (RP2D) | Up to 24 months
  The safe dose that demonstrates the greatest pharmacological activity.
PK evaluation of area under the plasma concentration versus time curve (AUC) of LP-118 | Up to Cycle 6 (each cycle is 28 days)
  AUC indicates the extent of exposure to LP-118 and its clearance rate from the body.
PK evaluation of peak plasma concentration (Cmax) of LP-118 | Up to Cycle 6 (each cycle is 28 days)
  Cmax indicates the highest drug concentration in the blood after LP-118 administration.
PK evaluation of time to maximum concentration (Tmax) of LP-118 | Up to Cycle 6 (each cycle is 28 days)
  Tmax indicates the time taken to reach the maximum drug concentration (i.e. Cmax).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  The proportion of patients who have a partial or complete response after LP-118 treatment.
Duration of response (DOR) | Up to 24 months
  The time from first documented response to disease progression or death.
Progression-free survival (PFS) | Up to 24 months
  The time from first dose to disease progression or death, whichever occurs first.
Overall survival | Up to 24 months
  The time from first dose to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Study Chair — Guangdong Provincial People's Hospital
Locations (4):
- China (4):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No